CLINICAL TRIAL: NCT04080960
Title: Dining With Diabetes in Pennsylvania
Acronym: DWD
Status: Completed | Type: Observational
Sponsor: Penn State University (Other)
Responsible Party: Sponsor
Other Study IDs: PRAMS00036501; 208113 (Other Grant/Funding Number: NNLM)
Record Dates: First submitted 2019-09-04; First posted 2019-09-06 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-06

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Lifestyle modification education — Lifestyle modification education and goal setting

SUMMARY:
Penn State Extension's Dining with Diabetes program is an evidence-based community education program for people with or at risk for type 2 diabetes. The program teaches participants how to prevent or manage their disease by providing practical knowledge and strategies to make the necessary lifestyle changes that will lead to healthier living and reduction in the risk of complications. The overall goals and objectives of the program are as follows:

Increasing knowledge of healthy food choices for families with or at risk for diabetes Promoting behavior changes by offering demonstrations and tasting of healthy food.

Increasing knowledge of essential medical tests associated with diabetes management.

Promoting physical activity as a component of diabetes control. Encouraging self-management and self-efficacy skill. Connecting participants to their healthcare providers for long-term follow-up. The program is designed to meet 4 consecutive weeks and then a 3 month follow-up. Participants A1c and blood pressure are taking at the first and follow-up classes. Classes consist of a nutrition lesson, physical activity, cooking demonstration and food tasting.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with type 2 diabetes individuals with pre-diabetes individuals at risk of developing type 2 diabetes healthy family members/caretakers healthy volunteers

Exclusion Criteria:

* under age 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults residents of Pennsylvania
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
hemoglobin A1C | 3 months
  participants can choose to have their hemoglobin A1C taken at the first and follow-up class, 3 months later

CONTACTS AND LOCATIONS:
Locations (1):
- Penn State University, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Griffie D, James L, Goetz S, Balotti B, Shr YH, Corbin M, Kelsey TW. Outcomes and Economic Benefits of Penn State Extension's Dining With Diabetes Program. Prev Chronic Dis. 2018 May 3;15:E50. doi: 10.5888/pcd15.170407. PMID 29729134